CLINICAL TRIAL: NCT03127436
Title: A Prospective, Open, Non-interventional Study to Assess the Tolerability and the Safety Profile of SCIT Therapy With Acarovac® Hausstaubmilbe in Patients With HDM-induced Rhinoconjunctivitis With or Without Allergic Asthma
Brief Title: Non-interventional Study to Assess the Tolerability and the Safety Profile of SCIT Therapy With Acarovac® Hausstaubmilbe
Status: Completed | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Collaborators: Bencard Allergie GmbH (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ralph Mösges, Prof. Dr. med. Ralph Mösges, University Hospital of Cologne
Other Study IDs: Acarovac AT
Record Dates: First submitted 2017-04-13; First posted 2017-04-25 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acarovac Hausstaubmilbe: This prospective open multi-centre non-interventional study was initiated to document the tolerability and the safety profile of the subcutaneous allergen-specific immunotherapy with Acarovac in house dust mite allergic patients (children and adults) in routine medical care.
  During the up-dosing phase with Acarovac, patients will receive 4 injections in 1-2 week intervals with increasing allergen amount up to the individual maximum tolerable dose. After reaching the individual maximum tolerable dose patients will receive one maintenance dose in a 4 - 8 week interval.
  Data on tolerability are documented by the physicians.
  Interventions: Drug: Acarovac

INTERVENTIONS:
Drug: Acarovac — House dust mite sensitized Patients receive increasing doses of subcutaneous immunotherapy with Acarovac. During the up-dosing phase, patients will receive 4 injections in 1-2 week intervals with increasing allergen amount up to the individual maximum tolerable dose. After reaching the individual maximum tolerable dose patients will receive one maintenance dose in a 4 - 8 week interval.

SUMMARY:
Non-interventional Study to Assess the Tolerability and the Safety Profile of SCIT therapy With Acarovac® Hausstaubmilbe

DETAILED DESCRIPTION:
This prospective open multi-centre non-interventional study was initiated to document the tolerability and the safety profile of the subcutaneous allergen-specific immunotherapy with Acarovac® in house dust mite allergic patients in routine medical care.

During the up-dosing phase with Acarovac®, patients will receive 4 injections in 1-2 week intervals with increasing allergen amount up to the individual maximum tolerable dose. After reaching the individual maximum tolerable dose patients will receive one maintenance dose in a 4 - 8 week interval.

Data on tolerability are documented by the physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the age of 5 years and older suffering from a house dust mite induced allergic rhinitis

Exclusion Criteria:

* Patients suffering from acute or chronic infections or inflammations
* Patients suffering from secondary modifications of the target organ with function impairment (emphysema, bronchiectasis)
* Patients suffering from severe and uncontrolled asthma
* Patients with a known severe autoimmune disease
* Patients with active malignant disease
* Patients requiring beta-blockers
* Patients having any contraindication for the use of adrenaline
* Patients with a hypersensitivity to the excipients of the drug

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults, adolescents and children from the age of 5 on, who suffer from perenial allergic rhinoconjunctivitis causued by house dust mites.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Numbers of treatment-related local and systemic reactions following SCIT administration | over the overall duration of the study
  Tolerability and safety will be assessed by the frequency and intensity of local reactions at the injection site (wheal size 5-10 cm, > 10 cm ) and systemic reactions (skin, airways, others) through study completion.
  The study covers the four injections of the up-dosing phase and one injection of the maintenance phase of the immunotherapy course.

SECONDARY OUTCOMES:
Safety and Tolerability - frequency and intensity of adverse events | over the overall duration of the study
  Frequency and intensity of adverse events
Safety and Tolerability - local reactions at injection site | over the overall duration of the study
  Frequency and intensity of local reactions at the injection site (wheal size 5-10 cm, > 10 cm )
Safety and Tolerability - Number of systemic reactions | over the overall duration of the study
  Frequency and intensity of systemic reactions
Changes in rhinoconjunctivitis score | baseline and 3-6 month, depending on the intervals between the injections and the applied up-dosing scheme
  The rhinoconjunctivitis score combines rhinitis symptom intensity and conjunctivitis symptom intensity and will be assessed retrospectively and after the course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kramer, Prof. Dr., Study Director — Bencard Allergie GmbH
Locations (1):
- Praxis für Lungenheilkunde, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No